CLINICAL TRIAL: NCT00169650
Title: Laparoscopic Pyeloplasty: A Registry and Database
Brief Title: Laparoscopic Pyeloplasty Registry and Database
Status: Completed | Type: Observational
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 03-048
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Ureteral Obstruction
Keywords: UPJ Obstruction; Renal Obstruction; Delayed Renal Flow
MeSH Terms: conditions — Ureteral Obstruction | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Registry and database of subjects undergoing laparoscopic pyeloplasty for ureteropelvic junction obstruction
  Interventions: Other: Registry and database

INTERVENTIONS:
Other: Registry and database — Subjects undergoing laparoscopic pyeloplasty for ureteropelvic junction obstruction at Methodist Urology in Indiana will be asked to participate in a registry and database to review outcomes of the surgery.

SUMMARY:
The gold standard for the treatment of ureteropelvic junction obstruction (UPJO) is the open pyeloplasty. As a minimally invasive alternative, many centers are currently offering laparoscopic pyeloplasty (LP) as primary therapy for UPJOs. Recent data has shown that laparoscopic pyeloplasty has comparable success rates to open pyeloplasties and produces durable results. The researchers are compiling a registry and database to review outcomes of laparoscopic pyeloplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of Methodist Urology in Indianapolis, IN over the age of 18 with ureteropelvic junction obstruction

Exclusion Criteria:

* Patients unable to give informed consent
* Patients with active bleeding diatheses
* Women who are pregnant or in whom pregnancy status cannot be confirmed
* Patients with medical conditions precluding laparoscopy
* Patients with active urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing laparoscopic pyeloplasty for ureteropelvic junction obstruction
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2003-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To record and review the surgical outcomes of our population of UPJO patients who have been treated with LP. Once all retrospective data has been reviewed, we will continue to collect outcome data on a prospective basis | One year

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States